CLINICAL TRIAL: NCT06254833
Title: Microdosing ICG for Serial Colonic Perfusion Study During Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanglei Liu (Other)
Responsible Party: Sponsor-Investigator, Shanglei Liu, Assistant Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 311249-00001
Record Dates: First submitted 2024-01-11; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Perfusion; Complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- regular dose ICG (No Intervention)
- micro dose icg (Active Comparator)
  Interventions: Other: micro dosing of ICG

INTERVENTIONS:
Other: micro dosing of ICG — smaller dose of injection of ICG. All devices used are FDA approved in clinical use.
  Other Names: small dose of injection if icg
  Arms: micro dose icg

SUMMARY:
using microdosing of ICG vs regular dosing of ICG for perfusion assessment during surgery

DETAILED DESCRIPTION:
Randomized dosing of 7.5mg or 0.75mg of ICG injection during surgery for bowel perfusion assessment using new imaging equipment

ELIGIBILITY:
Inclusion Criteria:

* all patient undergoing intestinal resection surgery

Exclusion Criteria:

* pregnancy, renal insufficiency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
ability to assess perfusion | up to 30 days post operatively
  likert scale evaluation survey performed by surgeon

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No